CLINICAL TRIAL: NCT02699632
Title: Research Participation in the Pregnant Population: A Survey Study
Brief Title: Participate While Pregnant Survey
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Leanne Redman, Principal Investigator, Pennington Biomedical Research Center
Other Study IDs: PBRC 2015-068
Record Dates: First submitted 2016-01-21; First posted 2016-03-04 (Estimated); Results first posted 2018-02-19 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-08

CONDITIONS: Pregnancy
Keywords: Survey

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The main goal for this study is to assess concerns and barriers to research participation by pregnant women through an anonymous online survey (www.pbrc.edu/ParticipateWhilePregnantSurvey).

DETAILED DESCRIPTION:
Participants will complete an online survey distributed through HIPAA compliant REDCap database. Collected data will consist of general multiple choice responses and optional "write-in" responses (e.g. providing a personal response for elaboration an "Other" option). No private health information will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Any individual may complete this survey.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited online. Anyone can take this survey, however females who have been pregnant or are planning to become pregnant will be the most relevant population.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leanne M Redman, PhD, MS, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sutton EF, Cain LE, Vallo PM, Redman LM. Strategies for Successful Recruitment of Pregnant Patients Into Clinical Trials. Obstet Gynecol. 2017 Mar;129(3):554-559. doi: 10.1097/AOG.0000000000001900. PMID 28178062

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: The survey was taken by 360 women previously, currently, or planning to become pregnant.
  Although number of unique site visitors between January and June 2016 is indeterminable, we had a completion rate of 69% (the percentage of surveys completed out of the total number initiated, ie, number of page 2 completions and number of page 1 completions).
Period: Overall Study
Arm/Group | All Participants
Started | 360
Completed | 358
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Women previously, currently, or planning to become pregnant. Data utilized is from completed questionnaires only, is uncorrected, and was collected from January through June 2016.
  Mode of initial contact with potential participants was made on the Internet (email and Facebook posts). Participants were instructed of survey length in these Internet advertisements and study purpose and data storage information on the first page of our electronic survey.
  No incentives were offered to participants, no protected health information was collected, and no measures were used for prevention of multiple entries from the same individual.
Arm/Group | All Participants
Number analyzed (Participants) | 360
Age, Customized [Count of Participants; unit: Participants]
  18-20 years | 3
  21-25 years | 42
  26-30 years | 123
  31-45 years | 182
  >45 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 360
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 47
  White | 286
  More than one race | 10
  Unknown or Not Reported | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 360

OUTCOME MEASURES:

1. Primary Outcome: Willingness to Participate in Research While Pregnant
Description: Survey question: What types of research would you be willing to participate in while you were pregnant?
Time Frame: Day 1
Population: part 1 of question observational studies; part 2 of question retrospective studies; part 3 of question lifestyle interventions in pregnancy
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: Respondents were asked what types of research they were willing to participate in during pregnancy
Arm/Group | All Participants
Number analyzed (Participants) | 358
Participants
  Observational Studies: Yes | 319
  Observational Studies: No | 39
  Retrospective Studies: Yes | 288
  Retrospective Studies: No | 70
  Lifestyle Interventions in Pregnancy: Yes | 308
  Lifestyle Interventions in Pregnancy: No | 50

2. Secondary Outcome: Preferred Methods for Learning About a Research Study
Description: Survey respondents were asked how they would prefer to learn about a research study with several answers cited.
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: Survey respondents were asked how they would prefer to learn about a research study
Arm/Group | All Participants
Number analyzed (Participants) | 358
Participants
  In person by my health care provider | 222
  in person by someone I didn't know | 130
  Other | 6

3. Secondary Outcome: Comfort of Participating in Research While Pregnant
Description: Survey question: Would you feel comfortable participating in a research study while pregnant?
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: Survey respondents were asked about their comfort and whether or not their physician needed to be involved.
Arm/Group | All Participants
Number analyzed (Participants) | 358
Participants
  Yes- if my physician approved | 222
  Other | 136

4. Secondary Outcome: Concerns for Participating in Research While Pregnant
Description: Survey question: What concerns might make you hesitant to participate in a research study while pregnant?
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: Survey respondents were asked about their concerns and what could be done to help minimize those concerns.
Arm/Group | All Participants
Number analyzed (Participants) | 358
Participants
  physician's approval would ease concerns | 233
  other | 125

ADVERSE EVENTS:
Description: Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Completeness checks were not used.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No